CLINICAL TRIAL: NCT00201188
Title: Cueing Patient-Clinician Collaboration to Improve Asthma
Brief Title: Enhancing Collaboration Between Doctors and Patients to Improve Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 279; R01HL073098 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2013-03-11 (Estimated); Status verified 2013-03

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive feedback and peak flow monitoring reports from their doctors.
  Interventions: Behavioral: Status Reports
- 2 (No Intervention): Participants will receive usual care.

INTERVENTIONS:
Behavioral: Status Reports — Interpreted Analysis of Peak-Flow Monitoring Trends
  Arms: 1

SUMMARY:
The purpose of this study is to improve anti-inflammatory medication adherence and asthma outcomes by using reports of peak flow monitoring to prompt communication between patients and their doctors.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is a chronic, potentially life-threatening disease that affects 17 million people in the United States. Asthma leads to millions of lost work days and thousands of hospitalizations annually. For the millions of people with this disease, it is chronic but controllable. Corticosteroids are the most effective medication for the long-term treatment of persistent asthma, and inhaling the medication minimizes the potential for systemic side effects. Despite convincing evidence of the benefits of inhaled corticosteroids (ICS), both patients and doctors seem reluctant to use them regularly. Many people who are prescribed ICS either never take them, or take them less frequently (e.g., once rather than twice daily), less regularly (e.g., "as needed" rather than daily), or at lower doses than prescribed. Doctors agree that at least 50% of people who are prescribed ICS fail to benefit fully because of poor adherence. The many reasons for non-adherence are not fully understood. The relationship between the doctor and patient, an area in which potential impact can be made, is believed to be the strongest predictor of medication adherence. Providing pertinent information about asthma related lung function should prompt communication between the patient and doctor to improve adherence to ICS.

DESIGN NARRATIVE:

The overall purpose of this study is to improve anti-inflammatory medication adherence and asthma outcomes by encouraging communication between patients and their doctor. The specific aims of the study include the following: 1) improve adherence to ICS medication by encouraging patient-doctor communication with feedback of objective information about airflow obstruction to reinforce medication-taking behavior; and 2) document the impact that the encouragement of communication has on health care outcomes, including health care utilization, pulmonary function, need for rescue courses of oral steroids, and functional impact. The hypothesis of the study is that informing patients and their primary care doctors about the degree of airflow obstruction will prompt interaction between them resulting in greater adherence to ICS medication over one year than will occur in a control group of similar patients who do not receive feedback. Promoting communication between adults with asthma and their doctors in a primary care clinical setting has not yet been studied. All doctors within three general medicine practices and their adult patients with moderate to severe asthma will be enrolled and assigned to either the intervention or usual care. Feedback of interpreted peak flow graphs in relation to current medication therapy will prompt the communication. The intent is to encourage and support the relationship between the doctor and patient rather than to directly intervene. The power of encouraging communication lies in the ensuing dialogue between the doctor and patient. Improvement of adherence to ICS among people with moderate or severe asthma has been shown to decrease morbidity of asthma and improve health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Asthma
* Currently using ICS
* Planning to live in the San Francisco Bay Area in the year following study entry

Exclusion Criteria:

* Diagnosis of any lung disease other than asthma
* Has a smoking history greater than or equal to 15 pack-years
* Psychological problems that may make monthly study visits impossible

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2003-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Adherence to ICS medication | Measured on a monthly basis

CONTACTS AND LOCATIONS:
Overall Officials: Susan L. Janson, DNSc,ANP,RN, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, Parnassus Campus, San Francisco, California, United States

REFERENCES:
- [Derived] Janson SL, McGrath KW, Covington JK, Baron RB, Lazarus SC. Objective airway monitoring improves asthma control in the cold and flu season: a cluster randomized trial. Chest. 2010 Nov;138(5):1148-55. doi: 10.1378/chest.09-2394. Epub 2010 Jun 10. PMID 20538819